CLINICAL TRIAL: NCT03281252
Title: A Prospective Study of Evaluation of Minor Bleeding and Utility of Bleeding Criteria in Acute-on-chronic Liver Failure Patients in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-07

CONDITIONS: Liver Failure, Acute on Chronic; Hemostatic Disorder
Keywords: liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hemostatic Disorders; Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ineffective hemostasis or a paradoxical prothrombotic state of Acute-on-chronic liver disease (ACLF) has been well established. However, the minor and major bleeding events has not been described yet. We observe the patients' major and minor bleeding events and use 4 criteria, which include BARC, ISTH, TIMI, Gusto ,to evaluate the incident rate of bleeding events in ACLF patients and pre-ACLF patients.

ELIGIBILITY:
Inclusion Criteria:

* patient with previously or undiagnosed chronic liver disease/cirrhosis;
* serum bilirubin higher than 3 mg/dl (51 mmol/L) or ALT>10ULN（male 300 U/L; female 200 U/L)

Exclusion Criteria:

* those who had or been diagnosed hepatocellular carcinoma or other types of malignancies;
* pregnancy;
* obstructive biliary diseases or other disease lead to bilirubin evaluation;
* using steroid or immunosuppressant in 4 weeks;
* prior surgeries including splenectomy，subtotal splenectomy and disconnection，liver transplantation.
* combine with other disease lead to organ failure including heart failure (NYHA IV),respiratory failure（PaO2<60mmHg),renal insufficiency(CKD 5) and conscious disturbance (GCS<8)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pre-acute-on-chronic liver failure and acute-on-chronic liver failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-16 (Actual); Primary Completion 2017-09-16 (Estimated); Study Completion 2017-09-16 (Estimated)

PRIMARY OUTCOMES:
28-day progression | 28-day
  progressed to EASL or APASL defined ACLF or death

SECONDARY OUTCOMES:
major bleeding event | 90-day
  major bleeding event happen
28-day mortality | 28-day
  death within 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China